CLINICAL TRIAL: NCT03872089
Title: Transient Thermal Behavior and Diabetic Foot
Acronym: PICOTE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL18_0371
Record Dates: First submitted 2019-02-22; First posted 2019-03-13 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Patients Type 1 and 2; Podologic Grade From 0 to 3
Keywords: Infrared Thermography; Diabetic foot; Six minutes walking test; Microcirculation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): Measurements of the temperature of the plantar arch by thermal imaging. Result analysis regarding podologic grade ( 0-1-2-3)
  Interventions: Other: Infrared Thermography

INTERVENTIONS:
Other: Infrared Thermography — Measurements of the temperature of the plantar arch by thermal imaging (Infrared Thermography)

SUMMARY:
In our study, the investigators propose to analyze the transient thermal responses taken at the level of the sole of the foot, following the application of a cold stimulus. By combining a spatio-temporal analysis of these temperature fields and a thermal modeling of the heat transfer in the thickness of the foot, the investigators want to highlight differences between healthy feet vs. pathological feet. Therefore, the investigators will determine the transient thermal responses at the level of the sole of the foot and correlate them with the podological grade.

DETAILED DESCRIPTION:
Both plants of the patient's feet will be observed by a thermal camera. Static observations (taking a single image), or dynamic (taking a series of images) of the foot, will be made. In the latter case, the observation will be done after a brisk walk of 6 min. The instruction given to patients will be to go the furthest in 3 min and then come back in 3 min, all while walking. The observation will be made by cameras without contact. These thermal cameras are non-invasive and non-ionizing, there is no risk related to their use. The camera will be placed on a tripod, a few tens of centimeters from the foot, and connected to a laptop (for the images acquisition). A wooden box, painted black, will be placed around both feet to protect the scene from parasitic thermal radiation that can disturb temperature variations. Foam will protect the skin / wood interface. Electric resistances, fixed on the box, will be placed in the field of vision of the thermal camera to guarantee the good treatment of the images. These resistors will never be in contact with the patient. The area filmed by the camera will be limited to the sole arch and, sometimes, the hand of patients to see if a thermal anomaly is also present on this member.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic subjects (type 1 and 2)
* age above 18 years old
* able to walk
* affiliate to insurance regimen

Exclusion Criteria:

* unable to stay motionless
* pregnancy
* subjects with feet wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Thermal signals measured on plantar foot | At the inclusion
  Determine the transient thermal responses at the plantar foot
Correlation with podologic grade | At the inclusion
  The classification of foot risk, mentioned in 2007 in the HAS report, is as follows ([HAS 2007]) Diabetic Foot Report http://www.has-sante.fr/portail/upload/docs/application/pdf/_foot_diabetic.pdf, 2007 :
  * Grade 0: absence of sensitive neuropathy Grade 1: isolated sensitive neuropathy
  * Grade 2: sensitive neuropathy associated with arteriopathy of the lower limbs and/or foot deformities
  * Grade 3: history(s) of foot ulceration (grade3a) and/or lower limb amputation (grade 3b)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Sultan, MD-PhD, Principal Investigator — Equipe Nutrition Diabete- CHU Lapeyronie- Montpellier
Locations (1):
- CHU Montpellier - Lapeyronie hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No